CLINICAL TRIAL: NCT04842708
Title: Evaluation of Anti-COVID 19 Pfizer Vaccination Effect on COVID 19 Detection Using Breath Analysis
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scentech Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Cov-2-SMC-V-2020
Record Dates: First submitted 2020-12-29; First posted 2021-04-13 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers that are not to be vaccinated against COVID19 (No Intervention): Healthy Volunteers that are not eligible to be vaccinated against COVID19
- Healthy Volunteers that are assigned to be vaccinated against COVID19 (Experimental): Healthy Volunteers that are eligible to be vaccinated against COVID19
  Interventions: Diagnostic Test: vaccination against COVID19

INTERVENTIONS:
Diagnostic Test: vaccination against COVID19 — subjects will undergo breath biopsy sampling before, 4-7 days post-first vaccination dose, and 7-10 days post-second vaccination dose.
  Arms: Healthy Volunteers that are assigned to be vaccinated against COVID19

SUMMARY:
The objective of this study will be to evaluate the effect of vaccination on breath VOC content.

By capturing and analyzing the breath of anti-COVID-19 vaccinated subjects during the period of antibody production, the investigators will determine and quantify all the compounds associated with the body reaction to the COVID-19 antigen.

DETAILED DESCRIPTION:
The objective of this study will be to evaluate the effect of vaccination on breath VOC content.

By capturing and analyzing the breath of anti-COVID-19 vaccinated subjects during the period of antibody production, the investigators will determine and quantify all the compounds associated with the body reaction to the COVID-19 antigen.

Rapidly growing serological evidence shows that IgM, IgG, and IgA antibodies against the S or N proteins evolve rapidly in the serum of asymptomatic as well as symptomatic COVID-19 patients within a week of infection or symptom onset and stay elevated with progressing disease.

Since the standard serology testing at Shamir Medical center tracks the presence of IgG only, those serologic tests will be conducted before and 48 hours following the second vaccination dose.

Nevertheless, since IgM antibodies are known to be produced by four to seven days following the first dose of vaccination, although IgM serology testing cannot be performed, the investigators are interested in sampling breath at this time range, in order for them to correlate it with the changes in the subjects' physiologic condition.

Since this is an unknown metabolic volatile compound mixture, the goal will be to identify compounds and quantify them with a high level of precision and subsequently correlate them with the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years at the time of consent
* Capable of understanding written and/or spoken language
* Able to provide informed consent
* Assigned to undergo anti-COVID-19 vaccination

Exclusion Criteria:

* Age under 18 years old
* Under guardianship or deprived of liberty
* Pregnant or lactating woman
* Not eligible for anti-COVID-19 vaccination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Association between breath VOCs and IgG in blood following second vaccination dose. | Through the study completion, up to 1 month.
  VOCs profile found in breath will be correlatated with IgG profile in blood.

SECONDARY OUTCOMES:
Association between VOCs profile and participants' clinical or demographic characteristics | Through the study completion, up to 1 month.
  Identify potential exhaled biomarkers association with participants' characteristics (age, gender, symptoms-severity, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No
IPD is not to be shared with other researchers.